CLINICAL TRIAL: NCT03700632
Title: A Randomized Clinical Trial of Part-time Patching Therapy on Improvement of Deviation Control in 3 to 8 Year-old Children With Intermittent Exotropia
Brief Title: Part-time Patch Therapy for Treatment of Intermittent Exotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9611257005
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Intervention Model Description: the experimental group will be treated with part time patch therapy and control group will be observed without any treatment.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: care provider, investigator and outcome assessor will be unaware the group of participants. because of the nature of study, patch therapy vs no treatment, masking of participant will not be possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patch therapy (Experimental): The eyes are alternatively patched for 2 hours a day in cases without a dominant eye while in cases with dominancy, the dominant eye is patched five days a week and the non-dominant eye is patched two days a week.
  Interventions: Other: patch therapy
- Control (No Intervention): no intervention will be done

INTERVENTIONS:
Other: patch therapy — The eyes are alternatively patched for 2 hours a day in cases without a dominant eye while in cases with dominancy, the dominant eye is patched five days a week and the non-dominant eye is patched two days a week
  Arms: patch therapy

SUMMARY:
Intermittent exotropia is the most common type of exotropia in children. Treatment options are surgical and non surgical. Nonsurgical management include Correction of refractive errors, Active orthoptic treatments, Prisms and Occlusion therapy. Benefits of patch therapy are limiting suppression, reducing the frequency and amplitude of the deviation, changing the nature of the deviation (from constant to intermittent exotropia or from intermittent exotropia to exophoria), however, there is a concern that occlusion of the eyes may cause fusion failure and worsen deviation control. According to a few number of studies and controversy among the results of investigations, the investigators designed this randomized clinical trial study to determine the effect of partial patch therapy on the deviation control of children with intermittent exotropia.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent distance exotropia or constant distance exotropia at least 15Δ and intermittent near exotropia or exophoria

Exclusion Criteria:

* No child's cooperation in evaluation of deviation control and regular visits for follow-up examinations
* Anisometropia more than 1.50 D, hypermetropia more than 3.50 D, and myopia more than 4.50 D on cyclorefraction
* History of previous treatments including eye occlusion, minus therapy, and strabismus surgery
* Any eye and systemic diseases other than strabismus including neurologic diseases and developmental delay.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-05-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
3-point scale Deviation Control | 3 months after treatment
  the ability of the child to control his/her deviation at far and near was assessed based on an office control 3-point scale : Children are categorized according to the office control 3-point scale into three control groups: good, fair, and poor.
  Good control: deviation occurs only during covering the eye and fusion is quickly established after removing the cover without blinking and re-fixation.
  Fair control: deviation occurs only during covering the eye and fusion is established after removing cover by blinking or re-fixation does happen.
  Poor control: deviation occurs spontaneously without covering and fusion hardly happens with too much effort and after a long time.
3-point scale Deviation Control | 6 months after treatent
  the ability of the child to control his/her deviation at far and near was assessed based on an office control 3-point scale : Children are categorized according to the office control 3-point scale into three control groups: good, fair, and poor.
  Good control: deviation occurs only during covering the eye and fusion is quickly established after removing the cover without blinking and re-fixation.
  Fair control: deviation occurs only during covering the eye and fusion is established after removing cover by blinking or re-fixation does happen.
  Poor control: deviation occurs spontaneously without covering and fusion hardly happens with too much effort and after a long time.
6-point scale Deviation Control | 3 months after treatment
  the ability of the child to control his/her deviation at far and near was assessed based on the office control 6-point scale: Children are classified according to the office control 6-point scale into six groups of 0 to 5.
  In this classification, exotropia is ranked after 30 seconds of observation: constant exotropia is ranked 5th, exotropia in more than 50% of the observing time is ranked 4th, and exotropia in less than 50% of the observing time is ranked 3rd. If exotropia is not seen in 30 seconds, the classification is made based on the speed of deviation control and fusion return 10 seconds after covering the eyes: back of fusion in more than 5 seconds is ranked 2nd, fusion return between 1 and 5 seconds ranked 1st, and fusion return in less than 1 second is ranked 0.

SECONDARY OUTCOMES:
Near stereopsis | at the time of enrollment, 3 month later and 6 month later
  Stereo acuity is measured at 40 cm using the Titmus test
Fusion | at the time of enrollment, 3 month later and 6 month later
  fusion at far & near are measured using the Worth 4-dot test. The Worth 4-dot test is used at 50 cm and 6 m for evaluating central and peripheral suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Reza Akbari, MD, Principal Investigator — Farabi Eye Research Center, Tehran University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu CB, Fan DS, Wong VW, Wong CY, Lam DS. Changing patterns of strabismus: a decade of experience in Hong Kong. Br J Ophthalmol. 2002 Aug;86(8):854-6. doi: 10.1136/bjo.86.8.854. PMID 12140202
- [Background] Multi-ethnic Pediatric Eye Disease Study Group. Prevalence of amblyopia and strabismus in African American and Hispanic children ages 6 to 72 months the multi-ethnic pediatric eye disease study. Ophthalmology. 2008 Jul;115(7):1229-1236.e1. doi: 10.1016/j.ophtha.2007.08.001. Epub 2007 Oct 22. PMID 17953989
- [Background] Vishnoi SK, Singh V, Mehra MK. Role of occlusion in treatment of intermittent exotropia. Indian J Ophthalmol. 1987 Jul-Aug;35(4):207-10. No abstract available. PMID 3506931
- [Background] Pediatric Eye Disease Investigator Group; Cotter SA, Mohney BG, Chandler DL, Holmes JM, Repka MX, Melia M, Wallace DK, Beck RW, Birch EE, Kraker RT, Tamkins SM, Miller AM, Sala NA, Glaser SR. A randomized trial comparing part-time patching with observation for children 3 to 10 years of age with intermittent exotropia. Ophthalmology. 2014 Dec;121(12):2299-310. doi: 10.1016/j.ophtha.2014.07.021. Epub 2014 Sep 16. PMID 25234012
- [Background] Spoor DK, Hiles DA. Occlusion therapy for exodeviations occurring in infants and young children. Ophthalmology. 1979 Dec;86(12):2152-7. doi: 10.1016/s0161-6420(79)35295-2. PMID 555806
- [Background] Freeman RS, Isenberg SJ. The use of part-time occlusion for early onset unilateral exotropia. J Pediatr Ophthalmol Strabismus. 1989 Mar-Apr;26(2):94-6. doi: 10.3928/0191-3913-19890301-14. PMID 2709283
- [Background] Chutter CP. Occlusion treatment of intermittent divergent strabismus. Am Orthopt J. 1977;27:80-4. No abstract available. PMID 900625
- [Background] IACOBUCCI I, HENDERSON JW. OCCLUSION IN THE PREOPERATIVE TREATMENT OF EXODEVIATIONS. Am Orthopt J. 1965;15:42-7. No abstract available. PMID 14274107
- [Background] Suh YW, Kim SH, Lee JY, Cho YA. Conversion of intermittent exotropia types subsequent to part-time occlusion therapy and its sustainability. Graefes Arch Clin Exp Ophthalmol. 2006 Jun;244(6):705-8. doi: 10.1007/s00417-005-0195-0. Epub 2006 Feb 4. PMID 16463040
- [Background] AlKahmous LS, Al-Saleh AA. Does occlusion therapy improve control in intermittent exotropia? Saudi J Ophthalmol. 2016 Oct-Dec;30(4):240-243. doi: 10.1016/j.sjopt.2016.07.004. Epub 2016 Jul 25. PMID 28003783
- [Background] Coffey B, Wick B, Cotter S, Scharre J, Horner D. Treatment options in intermittent exotropia: a critical appraisal. Optom Vis Sci. 1992 May;69(5):386-404. doi: 10.1097/00006324-199205000-00008. PMID 1594200
- [Background] Mohney BG, Holmes JM. An office-based scale for assessing control in intermittent exotropia. Strabismus. 2006 Sep;14(3):147-50. doi: 10.1080/09273970600894716. PMID 16950743
- [Derived] Akbari MR, Mehrpour M, Mirmohammadsadeghi A. The influence of alternate part-time patching on control of intermittent exotropia: a randomized clinical trial. Graefes Arch Clin Exp Ophthalmol. 2021 Jun;259(6):1625-1633. doi: 10.1007/s00417-020-05065-0. Epub 2021 Jan 7. PMID 33415357